CLINICAL TRIAL: NCT01741753
Title: Phase Ib Study of BKM120 Combined With Abiraterone Acetate for Docetaxel-pretreated, Castrate-resistant, Metastatic Prostate Cancer
Brief Title: BKM120+Abiraterone Acetate for Metastatic CRPC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to slow accrual the supllier of BKM120 asked we cease further enrollment.
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Glenn Bubley, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-121
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer
Keywords: Docetaxel Pretreated; Castrate Resistant; Metastatic
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — NVP-BKM120; abiraterone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): BKM120+Abiraterone+Prednisone
  Interventions: Drug: BKM120; Drug: Abiraterone; Drug: Prednisone

INTERVENTIONS:
Drug: BKM120 — Orally, every morning
Drug: Abiraterone — Orally, 1000 mg, every morning
Drug: Prednisone — Orally, 5 mg, every morning

SUMMARY:
This research study is a Phase I clinical trial. Phase I clinical trials test the safety of an investigational drug, in this case an investigational drug combined with standard drug therapy. Phase I studies also try to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is still being studied and taht research doctors are trying to find out more about it. It also means that the FDA has not approved the drug for use in patients, including people with your type of cancer.

BKM120 is a drug that inhibits the ability of tumors to grow and survive, which may lead to better outcomes in many types of cancer.

Abiraterone acetate is a drug that is approved for the treatment of prostate cancer, and works by inhibiting an enzyme found in prostate tumor tissue. While taking abiraterone acetate, individuals must also take a glucocorticoid such as prednisone.

Most patients with castrate-resistant prostate cancer will receive treatment with docetaxel, after which treatment with the combination of abiraterone and prednisone has been shown to be effective. Evidence has shown an interaction between the pathways through which BKM120 and abiraterone act on cancer. Therefore, it is thought that the treatment of castrate-resistant prostate cancer will be enhanced by combining BKM120 with abiraterone plus prednisone. The purpose of this study is to determine a safe dose for the combination of daily oral BKM120, abiraterone acetate, and prednisone in patients with castrate-resistant metastatic prostate cancer who have received prior treatment with docetaxel.

DETAILED DESCRIPTION:
You will undergo a screening process to determine if you are eligible to participate in this trial. This process will include the following procedures: Tumor Biopsy, including a bone marrow biopsy, which is used to determine the kinds of cancer cells in your tumor and a Physical Examination, including weight, blood pressure, heart rate, respiratory rate and body temperature.

Since we are looking for the highest dose of the study drug that can be administered safely without severe or unmanageable side effects in participants that have docetaxel resistant CRPC, not everyone who participates in this research study will receive the same dose of the study drug. The dose you get will depend on the number of participants who have been enrolled in the study before you and how well they have tolerated their doses.

If you take part in this research study, you will be given a study drug-dosing calendar for each treatment cycle. There will be a 14 day lead in phase of BKM120 alone to assess for toxicity from this agent. After the lead in phase, the standard dose of abiraterone and prednisone will be added to the BKM120 treatment regimen. Treatment cycles will last 4 weeks (28 days), during which time you will be taking the study drug in combination with the standard drug therapy once daily. Your time of participation in the study will be based on how well you tolerate the experimental drug. You could be participating in the study for a period of days, or years, depending on the course of your cancer.

During each treatment cycle, you will be required to return to see your research doctor for a study visit on Day 1 of each cycle. For Cycle 1, you will also need to return on Days 8, 15 and 22.

The following procedures will be performed and samples will be collected at 1 or more study visits: Evaluation of side effects, Vital sign measurement, Heart function tests, Neuropsychologic exams, Performance status assessment, Tumor biopsy, Assessment of tumor, Blood samples.

We would like to keep track of your medical condition for the rest of your life. We would like to do this by calling you on the telephone once a year to see how you are doing. Keeping in touch with you and checking your condition every year will help us look at the long-term effects of the research study. You will be required to return to see your research doctor for an end of study visit, which will take place 4-8 weeks after you undergo prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed CRPC with metastatic bone disease
* Castrate resistant disease
* Life expectancy of at least 6 months
* At least four weeks from previous treatment
* At least four weeks since any major surgery or radiation therapy
* Using highly effective contraception

Exclusion Criteria:

* Thromboembolism within past 6 months
* History of diabetes
* Prior therapy with abiraterone
* Prior therapy with PI3K inhibitor
* Alcohol or drug dependence currently or within past 6 months
* Contraindications to biopsy, such as bleeding disorders
* On anticoagulants such as warfarin or heparin
* Active malignancy other than skin cancer or superficial bladder cancer
* Untreated brain metastases
* Acute or chronic liver, renal disease or pancreatitis
* Mood disorders judged by the investigator to interfere with study participation
* Active cardiac disease or history of cardiac dysfunction
* Uncontrolled hypertension
* Known HIV, Hepatitis B or C
* Serious non-healing wound, ulcer or bone fracture
* Known or suspected allergy to BKM120, abiraterone or prednisone
* Impairment of GI function

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12-29 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Safety Profile and MTD for BKM120/Abiraterone/Prednisone | 2 years
  Determine the safety profile and MTD for the combination of BKM120 and abiraterone plus prednisone

SECONDARY OUTCOMES:
Duration of Response in Expansion Cohort | 2 years
  Determine duration time of response (time to progression) in the expansion cohort
Impact of PTEN Status on Response Rate/Duration | 2 years
  Assess the impact of PTEN status on response rate and duration of response

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Bubley, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth-Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- See also: Beth Israel Deaconess Medical Center Cancer Clinical Trials Office. — https://portal.bidmc.org/Intranets/Clinical/Cancer-Center/CancerClinicalTrial.aspx